CLINICAL TRIAL: NCT05090969
Title: Study of Febrile Syndromes After Tick Bite
Acronym: FebriTick
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7992
Record Dates: First submitted 2021-10-12; First posted 2021-10-25 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-10

CONDITIONS: Febrile Syndrome
Keywords: Febrile syndrome; Tick bite; Anaplasma phagocytophilum
MeSH Terms: conditions — Tick Bites

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Febrile syndromes after tick bites can be caused by different microorganisms: bacteria (B. miyamotoi, A. phagocytophilum, R. helvetica…), parasites (Babesia spp) and viruses (TBE virus). The clinical picture is not specific but complications may appear depending on the microorganism identified (thrombosis with N. mikurensis, meningoencephalitis with B. miyamotoi and the TBE virus). Thus, in order to provide appropriate treatment and monitoring, the infection should be documented.

ELIGIBILITY:
Inclusion criteria:

* Major subject (≥18 years old)
* Subject whose sample was sent to the bacteriology laboratory for research on Anaplasma phagocytophilum between 2009 and August 2020

Exclusion criteria:

* Subject having expressed his opposition to his medical data and biological resources not being reused for scientific research.
* Subject under guardianship or guardianship
* Subject under safeguard of justice

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Major subject whose sample was sent to the bacteriology laboratory for research on Anaplasma phagocytophilum between 2009 and August 2020
Sampling Method: Non-Probability Sample
Enrollment: 940 (Estimated)
Dates: Start 2020-11-30 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Retrospective search for the presence of an emerging pathogen in the cohort of patients with febrile syndrome after tick bite | Files analysed retrospectively from January 01, 2009 to August 31, 2020 will be examined]

CONTACTS AND LOCATIONS:
Overall Officials: Benoit JAULHAC, MD, PhD, Principal Investigator — Service Laboratoire de Bactériologie - Hôpitaux Universitaires de Strasbourg; Pierre BOYER, MD, Principal Investigator — Service Laboratoire de Bactériologie - Hôpitaux Universitaires de Strasbourg
Locations (1):
- Service Laboratoire de Bactériologie - Hôpitaux Universitaires de Strasbourg, Strasbourg, France